CLINICAL TRIAL: NCT04965428
Title: Fear-focused Self-Compassion Therapy for Young Breast Cancer Patients' Fear of Cancer Recurrence: Study Protocol of a Randomized Controlled Trial
Brief Title: Fear-focused Self-Compassion Therapy for Young Breast Cancer Patients' Fear of Cancer Recurrence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaanxi Normal University (Other)
Collaborators: Shaanxi Provincial Cancer Hospital (Other)
Responsible Party: Principal Investigator, Lei, Zhu, Associate Professor, Shaanxi Normal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Self-compassion FCR
Record Dates: First submitted 2021-06-19; First posted 2021-07-16 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Fear of Cancer Recurrence
Keywords: Fear of Cancer Recurrence; Self-compassion Therapy; RCT

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fear-focused Self-Compassion Therapy (Experimental): Experimental group receives group face-to-face Fear-focused Self-Compassion Therapy for eight weeks.
  Interventions: Behavioral: Fear-focused Self-Compassion Therapy
- Usual care (No Intervention): The no intervention group receives usual care supported by hospital or coming from elsewhere for eight weeks.

INTERVENTIONS:
Behavioral: Fear-focused Self-Compassion Therapy — The Fear-focused Self-Compassion Therapy will be delivered as a group format. The intervention consists of eight group face-to-face sessions (60-90 minute for each session) and will be delivered by three trained therapists for eight weeks (sessions are weekly). Each intervention group involves 10 patients.
  Arms: Fear-focused Self-Compassion Therapy

SUMMARY:
Few studies have tailored psychological intervention for fear of cancer recurrence (FCR) in young breast cancer patients, and the long-term efficacy of psychological intervention and its underlying mechanism are still unknown. To fill this knowledge gap, this protocol aims to evaluate the short-term and long-term effectiveness of Fear-focused Self-Compassion Therapy, as well as this therapy's psychological and physiological mechanisms in reducing severe FCR in young women with breast cancer.

This study will be a randomized controlled trial recruiting 160 Chinese young female breast cancer patients with severe FCR. Participants will be randomized to the Fear-focused Self-Compassion Therapy group or control group (1:1). Measurement will be completed at baseline (T0), immediately completing intervention (T1), after 3 months (T2), after 6 months (T3) and after 12 months (T4). Primary outcomes are FCR severity; secondary outcomes are self-compassion, neurophysiological data (i.e., salivary alpha amylase and heart rate variability), attentional bias for FCR, rumination, catastrophizing thinking, and psychological symptoms. The Fear-focused Self-Compassion Therapy is based on the theories of FCR development and self-compassion, and consists of eight-week face to face group sessions.

ELIGIBILITY:
Inclusion Criteria:

* (1) are diagnosed with breast cancer (including various cancer stages and subtypes);
* (2) are aged 18-45 years;
* (3) can sign written informed consent;
* (4) can read and write Chinese;
* (5) have severe FCR, with scores > 13 on the FCRI severity subscale.

Exclusion Criteria:

* (1) currently have psychiatric and psychological illness;
* (2) have other types of tumor;
* (3) had a previous cancer recurrence;
* (4) are participating another psychological intervention at the start of the study or during their eight-week therapy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Fear of cancer recurrence (FCR) | Baseline
  Fear of cancer recurrence will be assessed using 42-item Fear of Cancer Recurrence Inventory (FCRI). This questionnaire consists of seven subscales, with a total score representing one's levels of FCR. A score of 13 or higher on 9-item severe subscale (ranges from 0-36) indicates a clinical FCR.
Change from Baseline Fear of cancer recurrence (FCR) after immediately completing intervention | After immediately completing intervention
  Fear of cancer recurrence will be assessed using 42-item Fear of Cancer Recurrence Inventory (FCRI). This questionnaire consists of seven subscales, with a total score representing one's levels of FCR. A score of 13 or higher on 9-item severe subscale (ranges from 0-36) indicates a clinical FCR.
Change from Baseline Fear of cancer recurrence (FCR) at 3 months | Baseline to 3 months
  Fear of cancer recurrence will be assessed using 42-item Fear of Cancer Recurrence Inventory (FCRI). This questionnaire consists of seven subscales, with a total score representing one's levels of FCR. A score of 13 or higher on 9-item severe subscale (ranges from 0-36) indicates a clinical FCR.
Change from Baseline Fear of cancer recurrence (FCR) at 6 months | Baseline to 6 months
  Fear of cancer recurrence will be assessed using 42-item Fear of Cancer Recurrence Inventory (FCRI). This questionnaire consists of seven subscales, with a total score representing one's levels of FCR. A score of 13 or higher on 9-item severe subscale (ranges from 0-36) indicates a clinical FCR.
Change from Baseline Fear of cancer recurrence (FCR) at 12 months | Baseline to 12 months
  Fear of cancer recurrence will be assessed using 42-item Fear of Cancer Recurrence Inventory (FCRI). This questionnaire consists of seven subscales, with a total score representing one's levels of FCR. A score of 13 or higher on 9-item severe subscale (ranges from 0-36) indicates a clinical FCR.

SECONDARY OUTCOMES:
Self-compassion | Baseline, immediately completing intervention, baseline to 3 months, baseline to 6 months, baseline to 12 months.
  Self-compassion will be measured by using the 12-item Self-compassion Scale-Short Form (SCS-SF) consisting of six facets: self-kindness (2 items), self-judgement (2 items), common humanity (2 items), isolation (2 items), mindfulness (2 items) and over-identification (2 items) . Responses were rated on a five-point scale from 1 (almost never) to 5 (almost always).
Salivary alpha amylase | Baseline and immediately completing intervention
  The salivary alpha amylase activity will be measured by using a hand-held salivary alpha amylase monitor manufactured by Nipro (Osaka, Japan). This analyzer can automatically measure the salivary alpha amylase activity within one minute (about 30 seconds for saliva collection and 30 seconds for analyzing). Participants will be asked to brush teeth before measurement and not allowed to intake any food, beverage, tobacco or liquor within an hour.
Heart rate variability (HRV) | Baseline and immediately completing intervention
  The HRV will be measured by using signal detection and amplification system (Biopac ECG100C) of MP150-Biopac data acquisition system. The CardioBatch will be used to compute the HRV. Participants will be asked not to intake any stimulant (e.g., caffein, alcohol), or cannot do any strenuous activity within four hours before measurement.
Attentional bias for FCR | Baseline and immediately completing intervention
  Attentional bias for FCR will be assessed by conducting the dot-probe task, including 200 trials with the stimuli of cancer-related words and utilized in previous study. The dot-probe task will be presented on a laptop computer and run by using Matlab. At the beginning of each trial, a "+" will present for 500 milliseconds in the center of the screen. After that, a pair of word stimuli with a neutral word (e.g., apple) and a cancer-related word (e.g., chemotherapy) will be presented for 500 milliseconds on the left and right sides of screen. Then, the probe stimuli will be presented at the position where the word stimuli just appear. Once the probe stimuli appear, participants should press button of the keyboard as soon as possible. After that, the screen will present 500 milliseconds of blanking, and the next trial will start.
Rumination | Baseline and immediately completing intervention
  Rumination will be measured by using the 4-item Cognitive Emotion Regulation Questionnaire Rumination Subscale (CERQ-RS). Each item of CERQ-RS ranges from 1 to 5. A higher total score means more severe rumination.
Catastrophizing thinking | Baseline and immediately completing intervention
  Catastrophizing thinking will be measured by using the 4-item Cognitive Emotion Regulation Questionnaire Catastrophizing Subscale (CERQ-CS). Each item of CERQ-CS ranges from 1 to 5. A higher total score means more severe catastrophizing thinking.
Psychological symptoms | Baseline, immediately completing intervention, baseline to 3 months, baseline to 6 months, baseline to 12 months.
  Psychological symptoms will be measured by using Hospital Anxiety and Depression Scale (HADS). This 9-item questionnaire consisting of both anxiety subscale and depression subscale, rates on five-point (0-4) scales. The total score ranges from 0 to 36, and a higher total score means more severe depression and anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhu, PhD, Principal Investigator — Shaanxi Normal University; Juntao Yao, PhD, Study Director — Shaanxi Provincial Cancer Hospital
Locations (1):
- Shaanxi Provincial Cancer Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Wei L, Yang X, Sun S, Yu Y, Xie J, Zhao J, Wang X, Zhu L, Yao J. Fear-focused Self-compassion Therapy for young breast cancer patients' fear of cancer recurrence: Study protocol of a randomized controlled trial. Front Psychiatry. 2022 Sep 23;13:941459. doi: 10.3389/fpsyt.2022.941459. eCollection 2022. PMID 36213912